CLINICAL TRIAL: NCT04589546
Title: Does High-dose Vitamin B3 Supplementation Prevent Major Adverse Kidney Events During Septic Shock? A Multicenter Randomized Controlled Study
Brief Title: Does High-dose Vitamin B3 Supplementation Prevent Major Adverse Kidney Events During Septic Shock?
Acronym: VITAKI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Dieppe (Unknown); Centre Hospitalier d'Abbeville (Other); Centre Hospitalier de Laon (Unknown); University Hospital, Caen (Other); Centre Hospitalier de Cherbourg (Unknown); University Hospital, Rouen (Other); Centre Hospitalier de Roubaix (Other); Centre Hospitalier de Bethune (Network); Hôpital Saint Philibert, Lomme (Unknown); Tourcoing Hospital (Other); Centre Hospitalier de Valenciennes (Network); Centre Hospitalier Arras (Other); Centre Hospitalier de Lens (Other); Centre Hospitalier de Calais (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2020_843_0027
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury; Septic Shock; Nicotinamide; Mortality
Keywords: Acute Kidney Injury; Septic Shock; Nicotinamide
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin B3 (Experimental)
  Interventions: Drug: Nicotinamide treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: Nicotinamide treatment — Nicotinamide (500 mg) will be mixed in 50 ml of 0.9% saline and administered intravenously every 12 h for a total of 72 h.
  Arms: Vitamin B3
Drug: placebo treatment — For the placebo group, an identical volume of 0.9% saline will be administered in the same manner.
  Arms: Placebo

SUMMARY:
Sepsis is the most common cause of acute kidney injury (AKI) in critically ill patients and is associated with a high mortality rate. Currently there is no available specific treatment to prevent or treat AKI in this setting. Many experimental and clinical data suggest that Nicotinamide, a safe and inexpensive vitamin, could be effective to prevent major adverse kidney events during septic shock. The main objective of the study is to show the superiority of Nicotinamide supplementation compared to the placebo group, in patients with septic shock admitted to intensive care. A 15% reduction in the incidence of major renal adverse events at day 30 is expected in the "Nicotinamide" group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with septic shock defined as sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation.
* Written informed consent

Exclusion Criteria:

* Presence of inclusion criteria for more than 24 hours
* Immediate indication to start renal replacement therapy at the time of randomization: Hyperkalemia≥ 6.5 mmol /l, metabolic acidosis with pH <7.15 not controlled by medical treatment, diuretic resistant acute pulmonary edema or accumulation of a toxic requiring dialysis.
* Formal indication of Nicotinamide supplementation according to the attending physician (eg pellagra, undernutrition, severe alcoholism)
* Known severe chronic kidney disease (clearance <30 ml /min) in the last 3 months preceding the setic shock or kidney transplant recipient.
* Moribund patient (estimated survival less than 24 hours)
* Patient who are not expected to survive to day 30 due to terminal-stage disease (terminal respiratory or heart failure, Child C cirrhosis, uncontrolled cancer)
* Resuscitated cardiac arrest
* Pregnant or lactating
* Legal tutorship and guardianship
* Lack of social security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
proportion of patients meeting one or more criteria for MAKE30 | 3 years after study start
  MAKE30 is : in-hospital mortality, receipt of new RRT, or persistent renal dysfunction defined as a final inpatient serum creatinine value ≥2 time baseline serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No